CLINICAL TRIAL: NCT05437419
Title: A Phase 1, Randomized, Placebo-controlled, Double-blind, Multiple Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of Oral Doses of TCK-276 in Patients With Rheumatoid Arthritis
Brief Title: A Study to Investigate Safety, Tolerability, and PK of Oral Doses of TCK-276 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teijin America, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCK-276-102
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Multiple Ascending Dose; autoimmune disease; Disease modifying antirheumatic drugs (DMARD)
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): The patient will receive Dose A of TCK-276 or matching placebo orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
  Interventions: Drug: TCK-276; Drug: TCK-276 Placebo
- Cohort 2 (Experimental): The patient will receive Dose B of TCK-276 or matching placebo orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
  Interventions: Drug: TCK-276; Drug: TCK-276 Placebo
- Cohort 3 (Experimental): The patient will receive Dose C of TCK-276 or matching placebo orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
  Interventions: Drug: TCK-276; Drug: TCK-276 Placebo
- Cohort 4 (Experimental): The patient will receive Dose D of TCK-276 or matching placebo orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
  Interventions: Drug: TCK-276; Drug: TCK-276 Placebo

INTERVENTIONS:
Drug: TCK-276 — Patients will receive an oral dose of TCK-276 QD under fed conditions from Day 1 to Day 7.
  Other Names: Cyclin Dependent Kinase 4/6 (CDK 4/6) Inhibitor; TEI-T01276
Drug: TCK-276 Placebo — Patients will receive an oral dose of TCK-276 matching placebo QD under fed conditions from Day 1 to Day 7.
  Other Names: Placebo

SUMMARY:
The study is to evaluate the safety, tolerability, and pharmacokinetic (PK) of multiple orally administered TCK-276 in both males and females with Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
This is a Phase 1, multi-center, double-blind, randomized, placebo-controlled, multiple ascending dose (MAD) study.

The study will consist of a Screening Visit (Days -1 to Day 10), Treatment duration (up to 11 days) and a Follow-up/end of treatment (EOT) visit.

This MAD study will consist of 4 cohorts of 8 patients (6 active treatment and 2 matching placebo, or a 3:1 ratio), each receiving an oral dose of TCK-276 or matching placebo for 7 days (once daily (QD) under fed condition). The first cohort will be divided into 2 subgroups to implement the sentinel dosing approach.

The study duration is approximately 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA and meeting the 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for RA.
* Patients between the ages of 18 and 64 years, inclusive, at the Screening Visit.
* Female patient must be not pregnant, not breast feeding and one of the following conditions need to apply:

  1. Of non-childbearing potential based on documented surgical treatment or post-menopausal, meaning patient had spontaneous amenorrhea for at least 12 months without alternate medical cause prior to Screening Visit and follicle stimulating hormone (FSH) > 40 U/mL at the Screening Visit.
  2. Of childbearing potential and using a highly effective method of contraception and agrees to remain on a highly effective method from the time of signing the informed consent form (ICF) until 21 days after the last dose.
* Male patient must agree to stay abstinent or must use together with his female partner(s) a form of highly effective contraceptive (failure rate of < 1% per year) from the time of signing the ICF until up to 3 months after the last dose of the study drug.
* Nonsmokers (or other nicotine use) as determined by history and by negative urine cotinine concentration at the Screening Visit and at Admission.
* Body mass index (BMI) between 18.5 and 32.0 kg/m2, inclusive, at the Screening Visit.
* Patient is required to have completed a COVID-19 vaccine regimen within no more than 5 months prior to screening to be eligible for the study.
* Permitted concomitant medications for any reason, must be on a stable dose.
* Permitted medications include: anti-malarials; nonsteroidal anti-inflammatory drugs including selective cyclooxygenase-2 inhibitors at approved dosage, and low dose oral corticosteroids; methotrexate concomitantly with folic acid or folinic acid.

Exclusion Criteria:

* Female patients who are breastfeeding or have a positive urine pregnancy test.
* Patients who are unable to eat the prescribed meals during the stay at the site; vegetarian or vegan.
* Patient has a history of significant drug allergy.
* Patient has used a study drug, any prohibited medication(s), over-the-counter (OTC) medications, vitamins, dietary and herbal supplements.
* Patient has a history of active suicidal ideation, or any psychiatric disorders that will affect the patient's ability to participate in the study.
* Patient has a current or recent history of uncontrolled, clinically significant infectious, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Patient with any of the laboratory abnormalities as per reference.
* Patient has a history of alcohol and/or drug abuse within 24 weeks.
* Patient has positive results for drug testing and breath alcohol test.
* Regular consumption of alcohol within 6 months prior to the Screening Visit.
* Patient has positive test for hepatitis B surface antigen (HBsAg), anti-hepatitis B core (HBc) antibodies, hepatitis C virus (HCV) antibody, and/or human immunodeficiency virus (HIV) antibody at Screening Visit.
* Patient has QT interval corrected for heart rate (QTc) using Fridericia's correction (QTcF) > 450 ms for males or QTcF > 470 ms for females either at the Screening Visit or Admission, based on safety 12-lead electrocardiogram (ECG). Patient has Screening or Admission ECG with second- or third-degree atrioventricular block, bundle branch block, arrhythmia (but not sinus arrhythmia or supraventricular premature beats), or illegible QT interval.
* Patient has history or evidence of cardiopathy, acute coronary syndrome, hypertrophic cardiomyopathy, myocarditis or QT prolongation syndrome.
* Patient is unwilling to abstain from drinks and foods containing alcohol, grapefruit, or caffeine
* Patient has donated blood or experienced acute blood loss (including plasmapheresis) of greater than 500 mL within 90 days prior to the first dose of study drug.
* Patients with a known immunodeficiency disorder. Have a history of a major organ transplant or hematopoietic stem cell/marrow transplant.
* Patients with infections requiring treatment or hospitalization within 14 days prior to the Screening Visit, parenteral antimicrobial therapy within 60 days prior to the Screening Visit, infected joint prosthesis; history of herpes zoster, active herpes simplex, or herpes simplex on suppressive therapy.
* Patient has a chronic hepatic disease or hepatic impairment.
* Patient has a history of Mycobacterium tuberculosis or positive interferon gamma release assay for tuberculosis (IGRA-TB) or abnormal chest X-ray (for positive IGRA-TB patients).
* Patient has a history of any lymphoproliferative disorder.
* Patient has a history of COVID-19 unless fully recovered with no sequelae for 14 days.
* Patient who had a severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated).
* Patient who has recent exposure to someone who has COVID-19 symptoms or positive test result.
* Patient who has a positive reverse transcription polymerase chain reaction (RT-PCR) test for Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-CoV-2).
* Patient who has clinical signs and symptoms consistent with SARS-CoV-2 infection.
* Patients may not receive any live/attenuated vaccine from 30 days prior to the Screening Visit until Day 14 Follow-up Visit.
* COVID-19 vaccine should not be given 1 week prior to the Screening Visit.
* Patients with malignancy or history of malignancy except adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ. Previous treatment with total lymphoid irradiation.
* History of recurrent inflammatory joint disease other than RA or history of any other autoimmune rheumatic diseases other than Sjogren's syndrome.
* Major surgery within 30 days prior to the Screening Visit or patients with planned surgery.
* Patients who have an abnormal chest X-ray for interstitial lung disease (ILD) and/or patients with history of ILD.
* History of fainting or family history of sudden death.
* Patient has any disorder that would interfere with the absorption, distribution, metabolism or excretion of study drug.
* Patient has a history of deep vein thrombosis and/or pulmonary embolism.
* Patient has poor venous access.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana Zubkovskaya, Study Director — Medical Director
Locations (8):
- United States (8):
  - Orange County Research Center, Tustin, California
  - St. Jude Clinical Research, LLC, Doral, Florida
  - SouthCoast Research Center, Inc, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Clinical Site Partners, LLC dba CSP Orlando, Winter Park, Florida
  - SMS Clinical Research, LLC, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Proposals should be directed to clinical-trials-contact@teijinpo.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.

REFERENCES:
- [Derived] Tasaki D, Tsuruda K, Sun S, Tsumura Y, Asano S, Suzuki Y, Tsujimoto S, Miura D, Sato H. A double-blind, placebo-controlled, randomized multiple dose phase 1b trial of a CDK4/6 inhibitor, TCK-276, in patients with active rheumatoid arthritis. Rheumatology (Oxford). 2025 Mar 1;64(3):1036-1044. doi: 10.1093/rheumatology/keae357. PMID 39002122

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: The patient will receive 10 mg of TCK-276 orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
- Cohort 2: The patient will receive 25 mg of TCK-276 orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
- Cohort 3: The patient will receive 75 mg of TCK-276 orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
  .
- Cohort 4: The patient will receive 175 mg of TCK-276 orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
- Pooled Placebo Group: The patient will receive matching placebo for TCK-276 orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Pooled Placebo Group
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 3: The patient will receive 75 mg of TCK-276 orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
- Pooled Placebo Group: The patient will receive matching placebo orally from Day 1 to Day 7 (once daily (QD) under fed conditions).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Pooled Placebo Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 5 | 6 | 29
  Male | 0 | 0 | 0 | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 5 | 6 | 7 | 28
  Not Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 1 | 4
  White | 6 | 5 | 4 | 6 | 6 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 8 | 32
Height [Mean (Standard Deviation); unit: cm] | 163.5 (3.6472) | 163.03 (5.8745) | 160.167 (6.4936) | 165.533 (11.6610) | 164.878 (5.2737) | 163.515 (6.800)
Weight [Mean (Standard Deviation); unit: kg] | 74.950 (7.5688) | 73.252 (6.6383) | 75.102 (5.3800) | 80.678 (9.3768) | 73.829 (4.5924) | 75.454 (6.8510)
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.035 (2.5991) | 27.605 (2.6567) | 29.278 (1.3073) | 29.438 (1.5542) | 27.219 (2.2859) | 28.247 (2.2170)

OUTCOME MEASURES:

1. Primary Outcome: Number ot Participants With Treatment Emergent Adverse Events
Description: To evaluate the safety and tolerability of multiple oral doses of TCK-276 or placebo in patients with rheumatoid arthritis (RA)
Time Frame: 42 days (duration of study)
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Pooled Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 2 | 2 | 2 | 1 | 2

2. Secondary Outcome: Cmax: Plasma Concentrations of TCK-276 and TEI-W00595 (Metabolite)
Description: Cmax: Plasma Concentrations of TCK-276 and TEI-W00595 with time-concentration profile
Time Frame: Day 1 and Day 7
Population: One subject each from Cohorts 1 and 3 was excluded due to the occurrence of an event that met the definition of exclusion from the PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
ng/mL
  Cmax TCK-276 day 1 | 28.6 (22.4) | 60.6 (27.0) | 195 (146) | 417 (222)
  Cmax TCK-276 day 7 | 30.8 (13.4) | 61.4 (20.0) | 158 (76.1) | 402 (107)
  Cmax TEI-W00595 day 1 | 8.41 (4.98) | 28.7 (9.20) | 93.6 (90.2) | 176 (98.5)
  Cmax TEI-W00595 day 7 | 12.7 (4.55) | 30.3 (8.47) | 92.4 (60.3) | 161 (55.5)

3. Secondary Outcome: Tmax: Time of Maximum Plasma Concentration Determined Directly From the Concentration-time Profile
Description: To evaluate tmax as pharmacokinetic (PK) variables of TCK-276 and its metabolite in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
h
  TCK-276 Day 1 | 2 [1 to 12] | 3 [0.5 to 6] | 3 [0.75 to 12] | 1.75 [1 to 8]
  TCK-276 Day 7 | 2 [1.5 to 4] | 2.47 [1.5 to 4.08] | 2 [0.50 to 4.00] | 2.5 [1.00 to 4.00]
  TEI-W00595 Day 1 | 4 [2 to 12] | 4 [1 to 23.92] | 4 [0.75 to 12] | 3 [2 to 8]
  TEI-W00595 Day 7 | 4 [2 to 4] | 3.5 [2 to 15.93] | 3 [3 to 4] | 3 [2 to 4]

4. Secondary Outcome: t½: Terminal Elimination Half-life
Description: To evaluate t½ as PK variables of TCK-276 and its metabolite in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
h
  TCK-276 Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3
  TCK-276 Day 1 | 6.61 (2.53) | 4.49 (1.36) | 5.14 (0.937) | 7.13 (1.67)
  TCK-276 Day 7: number analyzed (Participants) | 5 | 6 | 4 | 6
  TCK-276 Day 7 | 13.6 (5.46) | 11.4 (6.15) | 13.6 (7.73) | 11.0 (4.39)
  TEI-W00595 Day 1: number analyzed (Participants) | 4 | 5 | 4 | 5
  TEI-W00595 Day 1 | 4.78 (0.716) | 5.15 (1.60) | 5.53 (1.27) | 5.49 (1.28)
  TEI-W00595 Day 7: number analyzed (Participants) | 5 | 4 | 5 | 6
  TEI-W00595 Day 7 | 9.10 (5.73) | 10.7 (6.42) | 12.8 (5.28) | 11.7 (4.69)

5. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-time Curve Over a Dosing Interval, Tau = 24 Hours
Description: To evaluate AUCtau as PK variables of TCK-276 and its metabolite in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
h*ng/mL
  TCK-276 Day 1: number analyzed (Participants) | 4 | 4 | 5 | 4
  TCK-276 Day 1 | 125 (20.3) | 341 (68.1) | 1150 (653) | 1530 (660)
  TCK-276 Day 7 | 172 (32.8) | 363 (48.6) | 1050 (520) | 2220 (542)
  TEI-W00595 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 6
  TEI-W00595 Day 1 | 70.3 (13.5) | 231 (65.4) | 890 (718) | 1270 (772)
  TEI-W00595 Day 7: number analyzed (Participants) | 5 | 4 | 5 | 6
  TEI-W00595 Day 7 | 91.2 (15.4) | 247 (59.1) | 788 (566) | 1200 (414)

6. Secondary Outcome: AUC0-inf: Area Under the Plasma Concentration Time Curve From Pre-dose (Time 0) Extrapolated to Infinite Time
Description: AUC0-inf:Area under the plasma concentration time curve from pre-dose (time 0) extrapolated to infinite time (Days 1 and 7)
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
h*ng/mL
  TCK-276 Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3
  TCK-276 Day 1 | 132 (23.6) | 390 (124) | 1230 (792) | 1830 (632)
  TCK-276 Day 7: number analyzed (Participants) | 5 | 6 | 4 | 6
  TCK-276 Day 7 | 205 (43.5) | 426 (94.0) | 1380 (802) | 2680 (789)
  TEI-W00595 Day 1: number analyzed (Participants) | 4 | 5 | 4 | 5
  TEI-W00595 Day 1 | 74.2 (14.2) | 246 (68.2) | 1010 (880) | 1590 (882)
  TEI-W00595 Day 7: number analyzed (Participants) | 5 | 4 | 5 | 6
  TEI-W00595 Day 7 | 105 (28.7) | 295 (87.6) | 1050 (752) | 1480 (586)

7. Secondary Outcome: Clearance (CL)/F: Apparent Total Body Clearance (Parent Only)
Description: To evaluate CL/F as PK variables of TCK-276 in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
L/h
  TCK-276 Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3
  TCK-276 Day 1 | 77.5 (14.0) | 68.9 (20.8) | 103 (102) | 103 (31.1)
  TCK-276 Day 7 | 59.5 (10.1) | 70.0 (9.62) | 102 (83.2) | 83.0 (21.0)

8. Secondary Outcome: Vz/F: Apparent Volume of Distribution Based on Terminal Phase (Parent Only)
Description: To evaluate Vz/F as PK variables of TCK-276 in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
L
  TCK-276 Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3
  TCK-276 Day 1 | 702 (175) | 457 (213) | 813 (877) | 1010 (221)
  TCK-276 Day 7: number analyzed (Participants) | 5 | 6 | 4 | 6
  TCK-276 Day 7 | 1150 (456) | 1150 (573) | 1510 (571) | 1280 (399)

9. Secondary Outcome: MRT0-inf: Mean Residence Time Extrapolated to Infinity
Description: To evaluate MRT0-inf as PK variables of TCK-276 and its metabolite in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
h
  TCK-276 Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3
  TCK-276 Day 1 | 7.65 (2.67) | 9.74 (5.36) | 7.56 (2.11) | 6.46 (0.479)
  TCK-276 Day 7: number analyzed (Participants) | 5 | 6 | 4 | 6
  TCK-276 Day 7 | 10.8 (1.42) | 11.3 (3.38) | 14.5 (6.71) | 11.4 (2.81)
  TEI-W00595 Day 1: number analyzed (Participants) | 4 | 5 | 4 | 5
  TEI-W00595 Day 1 | 9.09 (3.26) | 9.07 (2.40) | 9.66 (2.34) | 9.21 (3.14)
  TEI-W00595 Day 7: number analyzed (Participants) | 5 | 4 | 5 | 6
  TEI-W00595 Day 7 | 11.2 (2.25) | 12.2 (4.36) | 15.5 (5.96) | 12.9 (3.30)

10. Secondary Outcome: Racc (Cmax): Accumulation Ratio Based on Cmax
Description: Racc (Cmax) calculated as Cmax on Day 7/Cmax on Day 1.
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
Ratio
  TCK-276 Day 7 vs Day 1 | 1.72 (1.69) | 1.22 (0.736) | 1.19 (1.06) | 1.21 (0.725)
  TEI-W00595 Day 7 vs Day 1 | 1.85 (1.09) | 1.08 (0.242) | 1.26 (0.547) | 1.10 (0.463)

11. Secondary Outcome: Racc (AUCtau): Accumulation Ratio Based on AUCtau
Description: Racc (AUCtau) calculated as AUCtau on Day 7/AUCtau on Day 1. To evaluate Racc (AUCtau) as PK variables of TCK-276 and its metabolite in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
Ratio
  TCK-276 Day 7 vs Day 1: number analyzed (Participants) | 4 | 4 | 5 | 4
  TCK-276 Day 7 vs Day 1 | 1.37 (0.146) | 1.12 (0.286) | 0.960 (0.231) | 1.43 (0.288)
  TEI-W00595 Day 7 vs Day 1: number analyzed (Participants) | 4 | 3 | 5 | 6
  TEI-W00595 Day 7 vs Day 1 | 1.33 (0.170) | 1.07 (0.252) | 0.971 (0.256) | 1.13 (0.357)

12. Secondary Outcome: Metabolic Ratio (MR) for Cmax
Description: Molar metabolic ratio of Cmax calculated as (Cmax [metabolite] × molecular weight of parent)/(Cmax [parent] × molecular weight of metabolite).
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
Ratio
  Day 1 Metabolite vs Parent | 0.349 (0.166) | 0.499 (0.191) | 0.448 (0.190) | 0.403 (0.115)
  Day 7 Metabolite vs Parent | 0.412 (0.106) | 0.490 (0.115) | 0.537 (0.147) | 0.383 (0.0937)

13. Secondary Outcome: MR for Area Under the Plasma Concentration-time Curve (AUC)Tau
Description: Molar metabolic ratio of AUC calculated as (AUC [metabolite] × molecular weight of parent)/(AUC [parent] × molecular weight of metabolite). To evaluate MR AUC as PK variables of TCK-276 and its metabolite in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
Ratio
  Metabolite vs Parent Day 1: number analyzed (Participants) | 4 | 5 | 5 | 6
  Metabolite vs Parent Day 1 | 0.542 (0.0559) | 0.656 (0.102) | 0.669 (0.173) | 0.540 (0.0959)
  Metabolite vs Parent Day 7: number analyzed (Participants) | 5 | 4 | 5 | 6
  Metabolite vs Parent Day 7 | 0.514 (0.0489) | 0.658 (0.0759) | 0.675 (0.187) | 0.511 (0.0879)

14. Secondary Outcome: MR for Area Under the Plasma Concentration-time Curve (AUC)0-inf
Description: Molar metabolic ratio of AUC calculated as (AUC [metabolite] × molecular weight of parent)/(AUC [parent] × molecular weight of metabolite) 0-inf. To evaluate MR AUC 0-inf as PK variables of TCK-276 and its metabolite in patients with RA after multiple ascending dose (MAD) administration
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
Ratio
  Metabolite vs Parent Day 1: number analyzed (Participants) | 4 | 5 | 4 | 5
  Metabolite vs Parent Day 1 | 0.542 (0.0579) | 0.654 (0.0941) | 0.697 (0.200) | 0.567 (0.0942)
  Metabolite vs Parent Day 7: number analyzed (Participants) | 5 | 4 | 5 | 6
  Metabolite vs Parent Day 7 | 0.495 (0.0561) | 0.641 (0.0653) | 0.677 (0.184) | 0.519 (0.103)

15. Secondary Outcome: Ae 0-24: Amount of Study Drug Excreted Unchanged in the Urine (Days 1 and 7)
Description: Ae 0-24: Amount of study drug excreted unchanged in the urine (Days 1 and 7) over 24 hours
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
mg
  TCK-276 Day 1 | 0.194 (0.0847) | 0.529 (0.318) | 2.02 (1.19) | 2.04 (1.14)
  TCK-276 Day 7 | 0.203 (0.0847) | 1.68 (2.46) | 1.47 (0.537) | 2.07 (0.781)

16. Secondary Outcome: Fe 0-24: Percentage of Study Drug Excreted Unchanged in the Urine (Days 1 and 7)
Description: Fe 0-24: Percentage of study drug excreted unchanged in the urine (Days 1 and 7) over 24 hours
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of drug
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
percentage of drug
  TCK-276 Day 1 | 1.94 (0.847) | 2.11 (1.27) | 2.70 (1.58) | 1.17 (0.651)
  TCK-276 Day 7 | 2.03 (0.847) | 2.33 (1.67) | 1.96 (0.716) | 1.19 (0.446)

17. Secondary Outcome: Clearance Renal (CLr): Renal Clearance (Days 1 and 7)
Description: CLr: Renal clearance Day 1 and Day 7 (24 hours)
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
L/h
  TCK-276 Day 1: number analyzed (Participants) | 4 | 4 | 5 | 4
  TCK-276 Day 1 | 1.67 (0.442) | 1.89 (0.814) | 2.09 (1.09) | 0.985 (0.286)
  TCK-276 Day 7 | 1.15 (0.422) | 1.47 (1.02) | 1.41 (0.576) | 0.850 (0.351)

18. Secondary Outcome: Ae 0-72: Amount of Study Drug Excreted Unchanged in the Urine (Day 7)
Description: Ae 0-72: Amount of study drug excreted unchanged in the urine (Day 7) over a 72 hour period
Time Frame: Day 7 0-72 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
mg | 0.229 (0.0952) | 2.05 (3.28) | 1.61 (0.616) | 2.21 (0.868)

19. Secondary Outcome: Fe 0-72: Percentage of Study Drug Excreted Unchanged in the Urine
Description: Fe 0-72: Percentage of study drug excreted unchanged in the urine on Day 7 (72 hours)
Time Frame: Day 7 0-72 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of drug
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 6 | 5 | 6
percentage of drug | 2.29 (0.952) | 2.45 (1.70) | 2.15 (0.822) | 1.26 (0.496)

ADVERSE EVENTS:
Time Frame: Any adverse events (AEs) occurring after the subject signed the informed consent form (ICF) were collected and monitored throughout the study via safety assessments, observation, and subject reporting. Period of time included a 28 day screening period, a 10 day treatment period and a 4 day follow up period.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Pooled Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 2/6 | 1/6 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=6) | Pooled Placebo Group (N=8)
Sinus Tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT05437419/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT05437419/SAP_001.pdf